CLINICAL TRIAL: NCT06133205
Title: Efficacy of Abdominal Catgut Embedding Combined With Auricular Acupressure Therapy for Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH110-REC3-107
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Acupuncture

STUDY DESIGN:
Intervention Model Description: two groups, randomized, pre-post intervention study
Who Masked: Participant
Masking Description: Masking patients and statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): In both groups, catgut embedding using disposable single-strand surgical suture Polydioxanone threads was embedded to the following abdominal acupoints: ST-24 (Huaroumen), ST-25 (Tianshu), ST26 (Wailing), REN-12 (Zhongwan), REN-9 (Shuifen), REN-6 (Qihai), REN-4 (Guanyuan) as baseline treatment.
  Patients in this arm also received auricular acupressure using ear seeds (Vaccaria seeds) in the following auricular acupoints: Shen Men, Stomach, Endocrine. Those points were chosen due to function that are related to weight loss.
  Interventions: Other: Catgut Embedding at acupoints
- sham group (Sham Comparator): In both groups, catgut embedding using disposable single-strand surgical suture Polydioxanone threads was embedded to the following abdominal acupoints: ST-24 (Huaroumen), ST-25 (Tianshu), ST26 (Wailing), REN-12 (Zhongwan), REN-9 (Shuifen), REN-6 (Qihai), REN-4 (Guanyuan) as baseline treatment.
  Patients in this arm also received auricular acupressure using ear seeds (Vaccaria seeds) in the following auricular acupoints:Lung, Eye, Ear Apex. The points were selected as control points as there is no clear indication on their ability to contribute to weight loss.
  Interventions: Other: Catgut Embedding at acupoints

INTERVENTIONS:
Other: Catgut Embedding at acupoints — Supplemented by auricular point therapy, can increase the effect of catgut embedding therapy.

SUMMARY:
Objective: obesity is an important risk factor of chronic diseases, which not only threatens people's health, but also an important topic of public health. The purpose of this study is to define obesity according to the norms of the World Health Organization, and to explore whether combined weight loss methods have an impact on weight loss.

Methods:

In this study, Combined treatment of abdominal acupoint catgut embedding was combined with auricular pellet acupressure, The wire used for catgut embedding in the experiment was polydioxanone (PDO) 。 This experiment was divided into two groups: the experimental group A and the control group B 。 The reference measurement basis is the data obtained by "Inbody" instrument, including height and weight, body mass index (BMI), basic metallic rate (BMR), Body Fat Percentage BFP) , waist hip ratio and the data of total cholesterol (TC) and triglycerides (TG) obtained from biochemical blood examination, through the comparison before and after the test, we can judge whether the method of this test can achieve a certain degree of curative effect on weight loss.

DETAILED DESCRIPTION:
Objective: obesity is an important risk factor of chronic diseases, which not only threatens people's health, but also an important topic of public health. The purpose of this study is to define obesity according to the norms of the World Health Organization, and to explore whether combined weight loss methods have an impact on weight loss.

Methods:

In this study, This study is a random Single Blind Random Blind Trial conducted at Acupuncture and Moxibustion department of China Medical University hospital, Taichung city, Taiwan. The study involved 2 groups divided in 1:1 ratio to an intervention group and a control group. The study Combined treatment of abdominal acupoint catgut embedding was combined with auricular pellet acupressure, The wire used for catgut embedding in the experiment was polydioxanone (PDO) 。 This experiment was divided into two groups: the experimental group and the control group。The reference measurement basis is the data obtained by "Inbody" instrument, including height and weight, body mass index (BMI), basic metallic rate (BMR), Body Fat Percentage BFP), waist hip ratio and the data of total cholesterol (TC) and triglycerides (TG) obtained from biochemical blood examination, through the comparison before and after the test, we can judge whether the method of this test can achieve a certain degree of curative effect on weight loss.

ELIGIBILITY:
Inclusion Criteria:

A. Age 25 to 45 years old B. In line with the World Health Organization's BMI standard diagnosis ≥ 25 C. Waist circumference of men ≥90 cm or waist circumference of women ≥80 cm D. Body fat rate of men>25%, body fat rate of women>30% E. The above B, C, D can be included if they meet one of them F. Complete written informed consent

Exclusion Criteria:

* A. Pregnant, breastfeeding, menopausal women B. There are malignant tumors of the heart, liver and kidneys C. Diagnosed with mental illness D. Participated in another study within three months E. There are people who are taking diet pills

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
body weight | 12 weeks
  body weight in kilograms measured at inclusion and at 12 weeks measured by "InBody" body analysis instrument
BMI | 12 weeks
  Body mass index (BMI) measured at inclusion and at 12 weeks measured by "InBody" body analysis instrument
basal metabolic rate | 12 weeks
  basal metabolic rate measured at inclusion and at 12 weeks measured by "InBody" body analysis instrument
Body fat percentage | 12 weeks
  Body fat percentage measured at inclusion and at 12 weeks measured by "InBody" body analysis instrument

SECONDARY OUTCOMES:
Triglycerides | 12 weeks
  Triglycerides levels in blood measured by blood tests on inclusion and at 12 weeks
Total cholesterol | 12 weeks
  Total cholesterol levels in blood measured by blood tests on inclusion and at 12 weeks
WHOQOL | 12 weeks
  WHOQOL numerical assessment of quality of life, fill in the questionnaire before the first treatment.
Skeletal muscle weight | 12 weeks
  Skeletal muscle weight measured at inclusion and at 12 weeks measured by "InBody" body analysis instrument
waist hip ratio | 12 weeks
  waist hip ratio measured at inclusion and at 12 weeks measured by "InBody" body

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided